CLINICAL TRIAL: NCT05852652
Title: The Effect of Combination Between Cryolipolysis and Aerobic Exercise in Reducing Abdominal Adiposity in Obese Subjects
Brief Title: Combination of Cryolipolysis and Aerobic Exercise in Reducing Abdominal Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ebrahim Elsayed Mohamed, the principle investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cryolipolysis
Record Dates: First submitted 2023-04-23; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Abdominal Obesity
Keywords: cryolipolysis,low calorie diet and areobic exercise
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- cryolipolysis and aerobic exercise (Experimental): in this arm we combined between Three Max cool shaping Cryolipolysis device (ESM-8l00MO; EunSung global, Korea) was utilised. Vacuum controllable heads with cold temperatures ranging from (-10to 5)°C were adjusted according to each patient's tolerance, after careful patient sensation examination and vital sign evaluation before and after each session ,they got two sessions and walked from 30 to 60 minutes in nearby park.Two Cryolipolysis treatments totaling 45 minutes each were administered to each patient in the experimental group at the hypogastrium region, 5 cm below the umbilicus, using an anti-freezing membrane to prevent cold burn, in order to conduct the treatment
  Interventions: Device: cryolipolysis and aerobic exercise

INTERVENTIONS:
Device: cryolipolysis and aerobic exercise — the patients in this arm adjusted low calorie diet . According to the Recommended Dietary Intake (RDI), the low-calorie diet plan with three carefully calculated meals had a balanced macronutrient quantity of carbohydrate and protein, was low in fat, and was abundant in fruits, vegetables, and dietary fibres.
  they got two cryolipolysis sessions,one session in the month ,they got two sessions in two months,then took our outcome measures with walking 60 minutes in the park

SUMMARY:
The purpose of the study is To investigate the adding effect of Cryolipolysis to aerobic exercise with low caliorie diet on waist-to-hip ratio , ultrasonography, body mass index and skin fold of subcutaneous fat tissue in abdominal adiposity in obese subjects

DETAILED DESCRIPTION:
Obesity is a serious disease marked by an increase in body weight of at least 20% over the ideal weight due to an accumulation of body fat.

The prevalence of obesity has hit epidemic levels over the past few decades, and numerous obesity-related illnesses, including heart conditions, certain types of cancer, and diabetes, have risen concurrently. Weight loss through lifestyle modification, including a hypocaloric diet and/or increased physical exercise, along with behavioural techniques to support these changes, is the basis for treating or preventing these diseases through therapeutic intervention. Such methods rarely result in an obese person reaching a normal body weight because the typical weight reduction from lifestyle change is between 5 and 10% of baseline weight.

Recently, studies have used numerous devices, including cavitation, radiofrequency, cryolypolysis, and other many devices, according to the World Health Organization, to solve this issue.

The FDA has approved the cryolipolysis device for cutaneous cooling as well as a number of other uses. Cryolipolysis is a novel non-invasive technique for the selective reduction of fat cells with controlled, localised cooling.

Clinicians use the waist measurement and waist-to-hip ratio to assess abdominal obesity. These actions have a clear correlation to many vascular diseases, including atherosclerosis and the risk of developing acute coronary syndromes.

Typically, low-calorie diets are low in fat ( 30% of energy intake), high in carbohydrates (55-60% of total daily energy consumption), and energy-reduced (deficit of 2100-4200 kJ/d: ) minimum of 4200-5040 kJ/d for women and 5040- 5880 kJ/d for men) Due to the acutely high energy cost and ability to increase fat utilization, aerobic exercise is frequently recommended in conjunction with calorie restriction. Numerous studies examined the effects of modest caloric restriction alone or in combination with aerobic exercise.According to studies, a walk/jog programme enhanced body fat reduction compared to a group that only followed a diet.

There is a gap in the literature regarding combining cryolipolysis and aerobic exercise for losing weight, particularly abdominal adiposity, despite the fact that numerous studies have supported the efficacy of each on weight loss. Therefore, the goal of this research is to ascertain whether losing abdominal adiposity would be more successful when cryolipolysis and aerobic exercise were combined.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of the subjects range from (30-40)kg/m2
* subjects have abdominal adiposity

Exclusion Criteria:

* patients with liver and kidney diseases
* patients who have sensitivity to cold
* patients who have auto-immune disease
* patients after caesarean section
* impaired peripheral circulation
* Raynauds disease
* pregnant or lactating women within 6 months
* paroxysmal cold hemogobulinemia
* individuals who had metabolic derangement such as type 2 dibetes

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
the waist-to-hip ratio | 2 months
  by tape measurment
abdominal skin fold | 2 months
  by fat caliper
body mass index | 2 months
  by equation of world health organization
fat thickness | 2 months
  by ultrasonography

CONTACTS AND LOCATIONS:
Locations (1):
- Heba Ebrahim Elsayed Mohamed, Cairo, Egypt